CLINICAL TRIAL: NCT03913741
Title: Open Label Phase 1/2 Trial of Tisotumab Vedotin in Japanese Subjects With Advanced Solid Malignancies
Brief Title: A Trial of Tisotumab Vedotin in Japanese Subjects With Advanced Solid Malignancies
Acronym: innovaTV 206
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genmab (Industry)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCT1015-06; JapicCTI-194639 (Registry Identifier: JAPIC)
Record Dates: First submitted 2019-03-29; First posted 2019-04-12 (Actual); Last update posted 2022-06-23 (Actual); Status verified 2021-12

CONDITIONS: Solid Tumor
Keywords: tisotumab vedotin; cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — tisotumab vedotin

STUDY DESIGN:
Intervention Model Description: Single Group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental tisotumab vedotin (Experimental): Open label, single arm trial where tisotumab vedotin will be administered
  Interventions: Drug: tisotumab vedotin

INTERVENTIONS:
Drug: tisotumab vedotin — Tisotumab vedotin will be administered intravenously once every 21 days. The dose levels will be determined by the starting dose and the escalation steps taken in the trial

SUMMARY:
Open Label Phase 1/2 Trial of Tisotumab Vedotin in Japanese Subjects with Advanced Solid Malignancies

DETAILED DESCRIPTION:
Part 1 of this trial will determine the maximum tolerated dose (MTD) and/or the recommended Phase 2 dose (RP2D) and the safety profile of tisotumab vedotin in subjects with solid malignancies. Part 2 of this trial will enroll subjects with cervical cancer to provide further data on the safety, tolerability, PK and anti-tumor activity

ELIGIBILITY:
Inclusion Criteria (Main):

* PART 1 ONLY: Subjects with locally advanced or metastatic solid tumors, who have experienced disease progression while on standard therapy or are intolerant of, or not eligible for, standard therapy.
* PART 2 ONLY: Subjects with extra-pelvic metastatic or recurrent cervical cancer including squamous cell, adenocarcinoma or adenosquamous histology who have experienced disease progressed on standard of care chemotherapy in combination with bevacizumab, if eligible.

Patients must not have received more than 2 prior systemic treatment regimens for recurrent or metastatic cervical disease.

* Measurable disease according to RECIST v1.1
* Must be at least 20 years of age on the day of signing informed consent
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Is not pregnant, breastfeeding, or expecting to conceive children within the projected duration of the trial and for at least 6 months after the last trial treatment administration
* Women of childbearing potential must agree to use adequate contraception during and for 6 months after the last dose of trial treatment administration
* A man who is sexually active with a WOCBP and has not had a vasectomy must agree to use a barrier method of birth control (Part 1 only)
* Must provide signed informed consent before any trial-related activity is carried out.

Exclusion Criteria (Main):

* PART 2 ONLY: Clinically relevant bilateral hydronephrosis which cannot be alleviated by ureteral stents or percutaneous drainage.
* Known past or current coagulation defects leading to an increased risk of bleeding.
* Ongoing major bleeding.
* Has an active ocular surface disease at baseline. Subjects with prior history of cicatricial conjunctivitis are ineligible

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-02-27 (Actual); Primary Completion 2020-08-14 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
Dose Escalation and Dose Expansion: Incidence of drug-related Adverse Events (AEs) and Serious Adverse Events (SAEs) by CTCAE v5.0 [Safety] | Throughout the trial - until 90 days after last dose of tisotumab vedotin
Dose Escalation and Dose Expansion: Incidence of Dose Limiting Toxicities (DLTs), AEs, SAEs, adverse events leading to discontinuation, deaths and clinical laboratory test abnormalities [Tolerability] | Throughout the trial - until 90 days after last dose of tisotumab vedotin
Dose Escalation: maximum tolerated dose (MTD) and the recommended Phase 2 dose (RP2D) of tisotumab vedotin | Up to 21 days after the first dose of tisotumab vedotin (each cycle is 21 days)
Dose Escalation and Dose Expansion Pharmacokinetics of tisotumab vedotin: Maximum concentration (Cmax) after dosing | Up to approximately 42 days after initial dose of tisotumab vedotin
Dose Escalation and Dose Expansion Pharmacokinetics of tisotumab vedotin: Area under the plasma concentration-time curve from time 0 to the last measurable concentration (AUC(0-t)) | Up to approximately 42 days after initial dose of tisotumab vedotin
Dose Escalation and Dose Expansion Pharmacokinetics of tisotumab vedotin : Rate at which the drug is removed from the body (CL) | Up to approximately 42 days after initial dose of tisotumab vedotin
Dose Escalation and Dose Expansion Pharmacokinetics of tisotumab vedotin: Elimination half-life of the drug (T½) | Up to approximately 42 days after initial dose of tisotumab vedotin
Dose Escalation and Dose Expansion Pharmacokinetics of tisotumab vedotin: Time after dosing at which the maximum drug concentration was observed (Tmax) | Up to approximately 42 days after initial dose of tisotumab vedotin
Dose Escalation and Dose Expansion: Assess immunogenicity of tisotumab vedotin by measuring and assessing Anti-drug Antibody (ADA) | Throughout and at the end of trial (up to 90 days after last dose of tisotumab vedotin)
  Summarized by descriptive statistics by trial part and dose

SECONDARY OUTCOMES:
Dose Escalation and Dose Expansion: Evaluate antitumor activity of tisotumab vedotin by assessing Objective Response Rate (ORR) (based on RECIST 1.1) | Up to approximately 6 months after the first dose of tisotumab vedotin
  ORR defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR)
Dose Escalation and Dose Expansion: Evaluate antitumor activity of tisotumab vedotin by assessing Duration of Response (DOR) (based on RECIST 1.1) | Up to approximately 6 months after the first dose of tisotumab vedotin
  The DOR for a responder is defined as the time from the participant's initial objective response to the first date of either disease progression or death, whichever occurs first.
Dose Escalation and Dose Expansion: Evaluate antitumor activity of tisotumab vedotin by assessing Time to Response (TTR) (based on RECIST 1.1) | Up to approximately 6 months after the first dose of tisotumab vedotin
  TTR for a responder is defined as the time from the start of treatment with study drug to the first objective tumor response observed.

CONTACTS AND LOCATIONS:
Overall Officials: Keiichi Fujiwara, Professor, Principal Investigator — Saitama Medical University International Medical Center
Locations (8):
- Japan (8):
  - National Cancer Center Hosptial East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - NHO Hokkaido Cancer Center, Sapporo, Hokkaido
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saitama Medical University International Medical Center, Hidaka-shi, Saitama
  - Shizuoka Cancer Center, Sunto-gun, Shizuoka
  - National Cancer Center Hospital, Chūōku, Tokyo-To
  - Keio University Hospital, Shinjuku-ku, Tokyo-To

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Yonemori K, Kuboki Y, Hasegawa K, Iwata T, Kato H, Takehara K, Hirashima Y, Kato H, Passey C, Buchbjerg JK, Harris JR, Andreassen CM, Nicacio L, Soumaoro I, Fujiwara K. Tisotumab vedotin in Japanese patients with recurrent/metastatic cervical cancer: Results from the innovaTV 206 study. Cancer Sci. 2022 Aug;113(8):2788-2797. doi: 10.1111/cas.15443. Epub 2022 Jun 15. PMID 35633184